CLINICAL TRIAL: NCT04114981
Title: Phase III Trial of Post-Surgical Single Fraction Stereotactic Radiosurgery (SRS) Compared With Fractionated SRS for Resected Metastatic Brain Disease
Brief Title: Single Fraction Stereotactic Radiosurgery Compared With Fractionated Stereotactic Radiosurgery in Treating Patients With Resected Metastatic Brain Disease
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A071801; NCI-2019-02394 (Registry Identifier: NCI Clinical Trial Reporting Program); U10CA180821 (NIH)
Record Dates: First submitted 2019-10-02; First posted 2019-10-03 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Malignant Neoplasm in the Brain
MeSH Terms: conditions — Brain Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (SSRS) (Active Comparator): Patients undergo SSRS over 1 session.
  Interventions: Radiation: Single Fraction Stereotactic Radiosurgery; Procedure: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm II (FSRS) (Experimental): Patients undergo FSRS over 3 or 5 daily sessions.
  Interventions: Radiation: Fractionated Stereotactic Radiosurgery; Procedure: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Radiation: Single Fraction Stereotactic Radiosurgery — Undergo SSRS
  Other Names: Stereotactic Radiosurgery
  Arms: Arm I (SSRS)
Radiation: Fractionated Stereotactic Radiosurgery — Undergo FSRS
  Other Names: Stereotactic Radiosurgery
  Arms: Arm II (FSRS)
Procedure: Quality-of-Life Assessment — Ancillary studies
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase III trial studies how well single fraction stereotactic radiosurgery works compared with fractionated stereotactic radiosurgery in treating patients with cancer that has spread to the brain from other parts of the body and has been removed by surgery. Single fraction stereotactic radiosurgery is a specialized radiation therapy that delivers a single, high dose of radiation directly to the tumor and may cause less damage to normal tissue. Fractionated stereotactic radiosurgery delivers multiple, smaller doses of radiation therapy over time. This study may help doctors find out if fractionated stereotactic radiosurgery is better or worse than the usual approach with single fraction stereotactic radiosurgery.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To ascertain if time to surgical bed failure is increased with fractionated stereotactic radiosurgery (FSRS) compared to single-fraction stereotactic radiosurgery (SSRS) in patients with resected brain metastasis.

SECONDARY OBJECTIVES:

I. To ascertain if there is better emotional well-being at 9 months as assessed by the Functional Assessment of Cancer Therapy-Brain (FACT-BR) in patients with resected brain metastasis undergoing FSRS compared to SSRS (Primary quality of life [QOL] objective).

II. To ascertain whether there is improved overall survival in patients with resected brain metastases who undergo FSRS compared to patients who receive SSRS.

III. To ascertain in patients with resected brain metastases whether there is improved overall QOL as assessed by the FACT-BR and Linear Analog Self-Assessment (LASA) in patients who receive FSRS compared to patients who receive SSRS (Secondary QOL objective).

IV. To compare the functional independence in patients who receive FSRS to patients who receive SSRS.

V. To tabulate and descriptively compare the post-treatment adverse events associated with the interventions, including the potential impact of immunotherapy and targeted therapy.

VI. To compare rates of radiation necrosis at 12 months in patients who receive FSRS to patients who receive SSRS.

VII. To evaluate if there is any difference in central nervous system (CNS) failure patterns (local, distant brain failure, local leptomeningeal disease, widespread leptomeningeal disease) in patients who receive FSRS compared to patients who receive SSRS after resection of brain metastasis.

VIII. To ascertain in patients with resected brain metastases whether there is increased time to whole-brain radiotherapy (WBRT) in patients who receive FSRS compared to patients who receive SSRS.

IX. To determine in long-term survivors (patients who are alive more than 12 months from time of randomization) whether there is better emotional well-being and overall QOL as assessed by the FACT-BR and LASA in patients who receive FSRS to the surgical bed compared to patients who receive SSRS (Secondary QOL objective).

X. To assess for differences in CNS failure patterns (surgical, local, distant brain failure, leptomeningeal disease) as well as radiation necrosis rates as assessed by central review in patients who receive FSRS compared to patients who receive SSRS after resection of a brain metastasis.

XI. To ascertain in patients with resected brain metastases whether there is improved QOL as assessed by all other total and individual FACT-BR and LASA items and subscale values in patients who receive FSRS compared to patients who receive SSRS (Exploratory QOL objective).

XII. To determine in patients with resected brain metastases whether there is less cognitive progression in patients who receive FSRS to the surgical bed compared to patients who receive SSRS (Exploratory cognitive objective).

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients undergo SSRS over 1 session.

ARM II: Patients undergo FSRS over 3 or 5 daily sessions.

After completion of study, patients are followed up at 30 days, at 3, 6, 9, 12, 16, and 24 months, then every 6 months until 5 years from randomization.

ELIGIBILITY:
Inclusion Criteria:

PRE-REGISTRATION:

* Pathology from the resected brain metastasis must be consistent with a non-central nervous system primary site. Patients with or without active disease outside the nervous system are eligible (including patients with unknown primaries), as long as the pathology from the brain is consistent with a non-central nervous system primary site.
* Three or fewer (i.e. 0 to 3) unresected brain metastases (as defined on the post operative magnetic resonance imaging [MRI]) at the time of screening.

  o Note: Dural based metastases (e.g. commonly seen in breast cancer) are eligible.
* Unresected lesions must measure < 4.0 cm in maximal extent on the contrasted post-operative treatment MRI brain scan. The unresected lesions will be treated with SRS as outlined in the treatment section of the concept.

  o Note: The metastases size restriction does not apply to the resected brain metastasis.
* One brain metastasis must be completely (gross total resection) resected =< 30 days prior to pre-registration.

  o NOTE: May not have had resection of more than one brain metastasis.
* The resected brain metastasis must measure 2 cm or larger on the pre-operative MRI.
* Resection cavity must measure < 5.0 cm in maximal extent and the resection must be complete (gross total resection) on the post-operative MRI obtained =< 30 days prior to pre-registration.
* Karnofsky performance status of >= 60.
* For women of childbearing potential only, a negative urine or serum pregnancy test done =< 7 days prior to pre-registration is required.

  * Men and women of childbearing potential must be willing to employ adequate contraception throughout the study and for men for up to 3 months after completing treatment.
  * A female of childbearing potential is a sexually mature female who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months).
* Ability to complete an MRI of the head with contrast.
* The brain metastasis must be located > 5 mm of the optic chiasm; the brain metastasis must be located outside the brainstem (i.e. not inside the brainstem).
* Must not have any prior whole brain radiation therapy.
* Past radiosurgery to other lesions is allowed.

  o NOTE: The surgically resected lesion cannot be the same location treated in the past with radiosurgery (i.e. repeat radiosurgery to the same location/lesion is not allowed on this protocol).
* May not have primary germ cell tumor, small cell carcinoma, or lymphoma.
* No evidence of leptomeningeal metastasis (LMD).

  o NOTE: For the purposes of exclusion, LMD is a clinical diagnosis, defined as positive cerebrospinal fluid (CSF) cytology and/or equivocal radiologic or clinical evidence of leptomeningeal involvement. Patients with leptomeningeal symptoms in the setting of leptomeningeal enhancement by imaging (MRI) would be considered to have LMD even in the absence of positive CSF cytology, unless a parenchymal lesion can adequately explain the neurologic symptoms and/or signs. In contrast, an asymptomatic or minimally symptomatic patient with mild or nonspecific leptomeningeal enhancement (MRI) would not be considered to have LMD. In that patient, CSF sampling is not required to formally exclude LMD, but can be performed at the investigator's discretion based on level of clinical suspicion.
* Must be fluent in English, Spanish, or French.

REGISTRATION:

• Completion of all baseline electronic patient-reported outcome (ePRO) quality of life measures (or booklet quality of life measures) and Montreal Cognitive Assessment (MoCA).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2019-11-19 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Surgical bed recurrence-free survival (SB-RFS) | From the time of randomization up to 2 years post radiation
  Surgical bed control is defined as the absence of new nodular contrast enhancement in the surgical bed. In other words, a surgical bed recurrence-free survival (SB-RFS) event is defined as radiographic evidence of a new contrast-enhancing lesion (specifically any new progressive enhancing nodularity) at the site of the surgical resection. Will use a stratified log-rank test that compares and will report the median SB-RFS times between the single fraction stereotactic radiosurgery (SSRS) and fractionated stereotactic radiosurgery (FSRS) arms while adjusting for the stratification factors.

SECONDARY OUTCOMES:
Change in Functional Assessment of Cancer Therapy-Brain (FACT-BR) Emotional sub-scale score | At 9 months
  The average change from baseline to 9 months in the Functional Assessment of Cancer Therapy-Brain (FACT-BR) Emotional sub-scale will be compared between randomization arms.
Functional Assessment of Cancer Therapy-Brain (FACT-BR) total score | At 9 months
  The average change from baseline to 9 months in the Functional Assessment of Cancer Therapy-Brain (FACT-BR) total score will be compared between randomization arms.
Linear Analog Self-Assessment (LASA) overall quality of life | At 9 months
  The average change from baseline to 9 months in the Linear Analog Self-Assessment (LASA) overall total score will be compared between randomization arms.
Functional Assessment of Cancer Therapy-Brain (FACT-BR) Emotional sub-scale score for long-term survivors | At 12 months
  Long-term survivors defined as patients who are alive more than 12 months from time of randomization. The average change from baseline to 12 months in the Functional Assessment of Cancer Therapy-Brain (FACT-BR) Emotional sub-scale for the long-term survivors will be compared between randomization arms.
Functional Assessment of Cancer Therapy-Brain (FACT-BR) total score for long-term survivors | At 12 months
  Long-term survivors defined as patients who are alive more than 12 months from time of randomization. The average change from baseline to 12 months in the Functional Assessment of Cancer Therapy-Brain (FACT-BR) total score for the long-term survivors will be compared between randomization arms.
Linear Analog Self-Assessment (LASA) overall quality of life for long-term survivors | At 12 months
  Long-term survivors defined as patients who are alive more than 12 months from time of randomization. The average change from baseline to 9 months in the Linear Analog Self-Assessment (LASA) overall total score for the long-term survivors will be compared between randomization arms.
Karnofsky Performance Status (KPS) | Up to 24 months
  The duration of Karnofsky Performance Status (KPS) functional independence will be the time to when the KPS scores per patient decrease below their baseline level and will be compared between treatment arms by the logrank test. Median durations of KPS functional independence will be reported and compared between randomization arms.
Barthel Activities of Daily Living (ADL) Index | Up to 24 months
  The duration of Barthel Activities of Daily Living (ADL) functional independence will be the time to when the ADL scores per patient decrease below their baseline level and will be compared between treatment arms by the logrank test. Median durations of ADL functional independence will be reported and compared between randomization arms.
Karnofsky Performance Status (KPS) for long-term survivors | Up to 24 months
  Long-term survivors defined as patients who are alive more than 12 months from time of randomization. The duration of Karnofsky Performance Status (KPS) functional independence will be the time to when the KPS scores per patient decrease below their baseline level and will be compared between treatment arms by the logrank test. Median durations of KPS functional independence for long-term survivors will be reported and compared between randomization arms.
Barthel Activities of Daily Living (ADL) Index for long-term survivors | Up to 24 months
  Long-term survivors defined as patients who are alive more than 12 months from time of randomization. The duration of Barthel Activities of Daily Living (ADL) functional independence will be the time to when the ADL scores per patient decrease below their baseline level and will be compared between treatment arms by the logrank test. Median durations of ADL functional independence for long-term survivors will be reported and compared between randomization arms.
Overall survival | Up to 5 years
  Overall survival time will be compared between the treatment arms using a stratified log-rank test. If the proportional hazards assumption is violated, a restricted means analysis will be used to compare overall survival between the two treatment arms. Median survival times per treatment arms will be reported.
Incidence of adverse events | Up to 24 months
  The Common Terminology Criteria for Adverse Events version 5.0 will be used. The proportion of patients experiencing any adverse event will be compared between the two treatment arms using a chi-square (or Fisher's exact test, if more appropriate).
Proportion of patients with radiation necrosis | At 24 months
  The proportion of patients with radiation necrosis within 24 months from of starting treatment will be compared between the treatment arms with a chi-square test (or Fisher's exact test if more appropriate).
Time until whole-brain radiotherapy (WBRT) due to any reason (e.g. surgical bed recurrence, recurrence/progression at another central nervous system [CNS] site) | Up to 24 months
  Time until whole-brain radiotherapy (WBRT) will be compared between the treatment arms using a stratified log-rank test. Median time until WBRT per treatment arms will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Paul D. Brown, MD, Study Chair — Mayo Clinic
Locations (232):
- United States (223):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Anchorage Radiation Therapy Center, Anchorage, Alaska
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - Banner Thunderbird Medical Center, Glendale, Arizona
  - Banner-University Medical Center Phoenix, Phoenix, Arizona
  - Mayo Clinic Hospital in Arizona, Phoenix, Arizona
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - Mercy Hospital Fort Smith, Fort Smith, Arkansas
  - NEA Baptist Memorial Hospital and Fowler Family Cancer Center - Jonesboro, Jonesboro, Arkansas
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Los Angeles County-USC Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Epic Care Cyberknife Center, Walnut Creek, California
  - University of Colorado Hospital, Aurora, Colorado
  - UCHealth Memorial Hospital Central, Colorado Springs, Colorado
  - Yale University, New Haven, Connecticut
  - Helen F Graham Cancer Center, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - Boca Raton Regional Hospital, Boca Raton, Florida
  - Morton Plant Hospital, Clearwater, Florida
  - UM Sylvester Comprehensive Cancer Center at Coral Gables, Coral Gables, Florida
  - UM Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Walter Knox Memorial Hospital, Emmett, Idaho
  - Idaho Urologic Institute-Meridian, Meridian, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Cancer Clinic, Sandpoint, Idaho
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - SIH Cancer Institute, Carterville, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Northwestern University, Chicago, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Illinois CancerCare-Dixon, Dixon, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin Cancer Treatment Center, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - OSF Saint Francis Radiation Oncology at Peoria Cancer Center, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Southwest Illinois Health Services LLP, Swansea, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic - Ames, Ames, Iowa
  - McFarland Clinic - Boone, Boone, Iowa
  - McFarland Clinic - Trinity Cancer Center, Fort Dodge, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - McFarland Clinic - Jefferson, Jefferson, Iowa
  - McFarland Clinic - Marshalltown, Marshalltown, Iowa
  - University of Kansas Cancer Center, Kansas City, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - University of Kansas Hospital-Indian Creek Campus, Overland Park, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Woman's Hospital, Baton Rouge, Louisiana
  - Maine Medical Center- Scarborough Campus, Scarborough, Maine
  - MedStar Franklin Square Medical Center/Weinberg Cancer Institute, Baltimore, Maryland
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - McLaren Cancer Institute-Bay City, Bay City, Michigan
  - Saint Joseph Mercy Brighton, Brighton, Michigan
  - Saint Joseph Mercy Canton, Canton, Michigan
  - Saint Joseph Mercy Chelsea, Chelsea, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - McLaren Cancer Institute-Flint, Flint, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - Karmanos Cancer Institute at McLaren Greater Lansing, Lansing, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - McLaren Cancer Institute-Macomb, Mount Clemens, Michigan
  - Ascension Providence Hospitals - Novi, Novi, Michigan
  - McLaren Cancer Institute-Northern Michigan, Petoskey, Michigan
  - McLaren-Port Huron, Port Huron, Michigan
  - Ascension Saint Mary's Hospital, Saginaw, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Cambridge Medical Center, Cambridge, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Fairview Clinics and Surgery Center Maple Grove, Maple Grove, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - Monticello Cancer Center, Monticello, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - Fairview Northland Medical Center, Princeton, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Coborn Cancer Center at Saint Cloud Hospital, Saint Cloud, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Fairview Lakes Medical Center, Wyoming, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Saint Louis Cancer and Breast Institute-Ballwin, Ballwin, Missouri
  - Parkland Health Center-Bonne Terre, Bonne Terre, Missouri
  - Cox Cancer Center Branson, Branson, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - Parkland Health Center - Farmington, Farmington, Missouri
  - Capital Region Southwest Campus, Jefferson City, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri
  - University of Kansas Cancer Center at North Kansas City Hospital, North Kansas City, Missouri
  - Delbert Day Cancer Institute at PCRMC, Rolla, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Saint Louis Cancer and Breast Institute-South City, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - Missouri Baptist Outpatient Center-Sunset Hills, Sunset Hills, Missouri
  - Mercy Hospital Washington, Washington, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Community Medical Hospital, Missoula, Montana
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Community Medical Center, Toms River, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Glens Falls Hospital, Glens Falls, New York
  - Mount Sinai Chelsea, New York, New York
  - Mount Sinai West, New York, New York
  - Mount Sinai Hospital, New York, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Upstate Cancer Center Radiation Oncology at Oneida, Oneida, New York
  - University of Rochester, Rochester, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Novant Health Forsyth Medical Center, Winston-Salem, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Cincinnati Cancer Center-West Chester, West Chester, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Saint Alphonsus Medical Center-Baker City, Baker City, Oregon
  - Saint Alphonsus Medical Center-Ontario, Ontario, Oregon
  - Legacy Good Samaritan Hospital and Medical Center, Portland, Oregon
  - Northeast Radiation Oncology Center, Dunmore, Pennsylvania
  - Fox Chase Cancer Center Buckingham, Furlong, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Guthrie Medical Group PC-Robert Packer Hospital, Sayre, Pennsylvania
  - Saint Francis Cancer Center, Greenville, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - Lexington Medical Center, West Columbia, South Carolina
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Baptist Memorial Hospital and Cancer Center-Memphis, Memphis, Tennessee
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Memorial Hermann Texas Medical Center, Houston, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Inova Schar Cancer Institute, Fairfax, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - Northwest Wisconsin Cancer Center, Ashland, Wisconsin
  - Ascension Southeast Wisconsin Hospital - Elmbrook Campus, Brookfield, Wisconsin
  - Ascension Saint Francis - Reiman Cancer Center, Franklin, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - University of Wisconsin Carbone Cancer Center, Madison, Wisconsin
  - Ascension Columbia Saint Mary's Hospital - Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Ascension All Saints Hospital, Racine, Wisconsin
  - UW Cancer Center at ProHealth Care, Waukesha, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Billings Clinic-Cody, Cody, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming
- Canada (9):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - University Health Network-Princess Margaret Hospital, Toronto, Ontario
  - CHUM - Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - The Research Institute of the McGill University Health Centre (MUHC), Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec
  - CHU de Quebec-L'Hotel-Dieu de Quebec (HDQ), Québec, Quebec
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: Yes